CLINICAL TRIAL: NCT00516555
Title: Ebis: The Eindhoven Breech Intervention Study
Status: Completed | Type: Observational
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Collaborators: Tilburg University (Other)
Responsible Party: Principal Investigator, S.Kuppens, MD, Phd, Catharina Ziekenhuis Eindhoven
Other Study IDs: M06/1130; ABR Number 14584
Record Dates: First submitted 2007-08-13; First posted 2007-08-15 (Estimated); Last update posted 2013-03-19 (Estimated); Status verified 2013-03

CONDITIONS: Breech Presentation; External Cephalic Version; Thyroid Hormones; Stress, Psychological; Congenital Hip Dysplasia
Keywords: Breech Presentation; External Cephalic version; Thyroid Function Tests
MeSH Terms: conditions — Breech Presentation; Stress, Psychological; Hip Dislocation, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples for thyroid hormone status (Tsh, Ft4, anti-TPO)
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- A, 07, 001: Pregnant women at term with a baby in breech presentation who will have an external cephalic version.

SUMMARY:
The purpose of this study is to evaluate whether successful external cephalic version is associated with maternal thyroid function and mood state in pregnant women with breech presentation at term.

The relationship between successful external cephalic version and neonatal thyroid function will also be investigated.

A possible beneficial effect of successful external cephalic version on the development of congenital hip dysplasia will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Single pregnancy
* Gestation of 35 weeks or more
* Appropriate knowledge of the Dutch language
* Fetus in any of the 4 types of breech presentation: frank breech, complete breech, incomplete breech or footling presentation

Exclusion Criteria:

* Previous caesarean section
* Indication for caesarean delivery irrespective of presentation
* Previous abruptio placenta
* Multiple pregnancy
* Ruptured membranes
* Non-reassuring fetal monitoring tests results
* Hyperextended fetal head
* Significant uterine or fetal anomaly
* Use of thyroid medication
* Maternal autoimmune disease (such as insulin-dependant diabetes mellitus)
* Intra-uterine growth retardation
* Oligohydramnios
* HIV-positive women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women with breech presentation at term in the region of Eindhoven, The Netherlands.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2007-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
The relation between maternal mood state and thyroid function during end gestation and successful external version of fetal breech position | during external cephalic version

SECONDARY OUTCOMES:
the relation between neonatal thyroid parameters at delivery and successful external version, the effect of successful version on hipdysplasia | at the time of delivery, at the age of 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Simone M. Kuppens, MD, Principal Investigator — Catharina Ziekenhuis Eindhoven; Tom H. Hasaart, MD, PhD, Study Director — Catharina Ziekenhuis Eindhoven; Victor J. Pop, MD, PhD, Prof, Study Chair — Tilburg University; H. Vader, PhD, Prof, Study Chair — Maxima Medisch Centrum Veldhoven
Locations (1):
- S.Kuppens, Eindhoven, North Brabant, Netherlands

REFERENCES:
- [Derived] Kuppens SM, Smailbegovic I, Houterman S, de Leeuw I, Hasaart TH. Fetal heart rate abnormalities during and after external cephalic version: Which fetuses are at risk and how are they delivered? BMC Pregnancy Childbirth. 2017 Oct 17;17(1):363. doi: 10.1186/s12884-017-1547-6. PMID 29041923
- [Derived] Ciliacus E, van der Zalm M, Truijens SE, Hasaart TH, Pop VJ, Kuppens SM. Fear for external cephalic version and depression: predictors of successful external cephalic version for breech presentation at term? BMC Pregnancy Childbirth. 2014 Mar 12;14:101. doi: 10.1186/1471-2393-14-101. PMID 24620740
- [Derived] Kuppens SM, Kooistra L, Hasaart TH, van der Donk RW, Vader HL, Oei GS, Pop VJ. Maternal thyroid function and the outcome of external cephalic version: a prospective cohort study. BMC Pregnancy Childbirth. 2011 Jan 26;11:10. doi: 10.1186/1471-2393-11-10. PMID 21269431